CLINICAL TRIAL: NCT01311817
Title: Transcutaneous Immunization With actA/plcB-Deleted Listeria Monocytogenes Expressing Influenza A Nucleoprotein (BMB72) and Cholera Toxin Adjuvant
Brief Title: Transcutaneous Immunization With an Attenuated Listeria Monocytogenes Vector Vaccine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Elizabeth L. Hohmann, MD, Associate Professor, Massachusetts General Hospital
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: 2008P-0002296
Record Dates: First submitted 2011-03-08; First posted 2011-03-10 (Estimated); Last update posted 2015-10-02 (Estimated); Status verified 2015-09

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Saline Patch (Placebo Comparator): 1mL saline applied to the vaccine patch
  Interventions: Biological: BMB72 (actA/plcB-deleted Listeria monocytogenes expressing influenza A nucleoprotein)
- Bacteria plus CT (Experimental): 0.95mL bacterial vector plus 0.05mL cholera toxin
  Interventions: Biological: BMB72 (actA/plcB-deleted Listeria monocytogenes expressing influenza A nucleoprotein)

INTERVENTIONS:
Biological: BMB72 (actA/plcB-deleted Listeria monocytogenes expressing influenza A nucleoprotein) — 1mL liquid contained in an adhesive skin patch
  Other Names: Lot ELH072910

SUMMARY:
This project is a pilot safety and immunogenicity study of transcutaneous vaccination with live attenuated Listeria monocytogenes BMB72 bacteria (actA/plcB-deleted, expressing influenza A nucleoprotein) and a cutaneous adjuvant, native purified cholera toxin. Transcutaneous vaccination is needle-less application of materials directly to the skin. Healthy adult volunteers (4 per group) will receive either:

* Saline (placebo)
* Cholera toxin adjuvant alone
* L. monocytogenes BMB72 bacteria alone
* L. monocytogenes BMB72 bacteria plus Cholera toxin adjuvant

Vaccine solutions will be applied to the upper deltoid area under a standard Tegaderm dressing. Key primary endpoints include: safety as measured primarily by clinical findings (VS, cutaneous exams, and systemic reactions), and immune responses as measured by serological responses to L. monocytogenes, influenza A nucleoprotein, CT, and IFN gamma ELISPOT responses to listeriolysin and nucleoprotein peptides. Local skin immune responses will be evaluated by skin biopsy in subjects who agree to that (optional). The study will begin with 2 "roll-in" subjects receiving both L. monocytogenes and CT.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult 18-55 years old, male or female.
* Adequate venous access by inspection for frequent blood draws.
* Must have normal physical exam and laboratory values within the normal range for age/gender in screening studies (see details below).
* Be willing to return for 3 vaccinations, and the needed follow-up visits.
* Not pregnant (WOCBP have pregnancy testing prior to vaccination, on a standard schedule over the course of the study, and must use contraception).
* Non-smokers (altered immunity).
* Body mass index (BMI) less than or equal to 32.5 (the obese have impaired responses to some vaccines).
* Normal skin exam.
* Volunteers must be feeling well and be afebrile (T<99.5) at the time of vaccination.

Exclusion Criteria:

* History of allergy to any penicillin (including penicillin G, penicillin V, ampicillin, amoxicillin) or sulfa drugs (trimethoprim/sulfamethoxazole is the second line agent for therapy of listeriosis).
* Any chronic medical illness or problem requiring chronic medical care. Exceptions:

  * Subjects on one antihypertensive prescribed for essential hypertension, with seated BP in the normal range at screening will be accepted. These are immunologically normal adults and we do not believe treated essential hypertension as a single illness puts these individuals at any greater risk than other healthy adults.
  * Subjects using only PRN beta agonists for mild asthma, or cold or exercise-induced bronchospams, will be allowed (those with any prior or current inhaled or systemic steroids for asthma are excluded).
* Any chronic or current skin disorder, e.g. eczema, dermatitis, psoriasis, rosacea, or acne. Prescription medications more than 5 years ago for teenage acne without current acne on exam or current use of those medications does not exclude subjects.
* Any acute skin break or problem at the planned vaccination site (deltoid).
* Upper extremity lymphedema, deformity (e.g. large burn or poorly-healed fracture), swelling or vascular abnormality on exam. A history of a distant isolated arm, wrist or hand fracture (more than 5 years earlier) with no residual functional deficit or visible deformity will not exclude a subject.
* History of allergy to medical bandages, tape, or adhesives (a Tegaderm patch is used for application.)
* No history of bleeding disorder, or anticoagulant medications. (The protocol has an optional skin biopsy).
* Pregnancy, attempting pregnancy, or unwillingness to use medically acceptable contraception for entire study period if sexually active. Women of childbearing potential will have serum pregnancy testing. Women who are menopausal (over 50 years of age with no menses for more than one year) or surgically sterilized are not considered of child-bearing potential and will not require pregnancy testing or contraception. Acceptable contraception includes: condoms/spermicide, prescription hormonal contraceptive pills, patches, rings, and implants; IUDs.
* Any type of chronic prescription medication use for any reason, including acne or skin conditions. Exceptions: oral contraceptives, depo contraceptives, patch contraceptives, one antihypertensive agent is allowed, if BP is normal on exam as noted above.
* History of keloid scars, or poor wound healing.
* Previous splenectomy or abdominal procedure where splenectomy was possibly performed - e.g. laparotomy for trauma. (Not a known risk factor for listeriosis, but might conceivably result in more serious illness, or alter immune responses to a bacterial pathogen).
* Any biomedical implants: cranial plates, joint prostheses, bone screws, pacemakers, CNS clips, and heart valves. (Exceptions: K wires or 3 or fewer dental implants more than 2 years post implantation in an otherwise healthy individual with no functional deficit or deformity will not exclude an individual.)
* Mitral valve click or prolapse or heart murmur beyond a typical flow murmur.
* Chronic pain syndromes like headaches or back pain requiring use (more than once per week) of over-the-counter medications like Tylenol or NSAIDs.
* Elevated iron stores, evidence of chronic hemolysis such as abnormal blood smear, elevated transferrin or transferrin saturation >50% (Iron overload predisposes to listeriosis and asymptomatic elevated iron level may indicate early iron overload state, i.e. hemochromatosis).
* Any evidence of immunosuppressive illness (e.g. HIV or malignancy) or seropositive for HIV or hepatitis B (sAg positive) or C, or history of frequent infections especially sino-pulmonary, skin or soft tissue or GI infections. Hepatitis B serologies consistent with vaccination or resolved prior infection (surface antibody positive and surface antigen negative) is not a reason for exclusion.
* Subjects who live with immunosuppressed individuals, children under 4 years of age, or people with chronic skin disorders in the household are excluded.
* Alcohol or substance abuse (immunosuppressive affects of alcohol and altered immune responses) by history. Occasional recreational use of marijuana, or social alcohol use are not exclusion criteria. Drug testing is not performed.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2011-01; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Vaccine Safety | 1 year +/-
  Safety is measured primarily by clinical findings (VS, cutaneous exams, and systemic reactions
Immunogenicity | 1 year +/-
  Immune responses are measured by serological responses to L. monocytogenes, influenza A nucleoprotein, cholera toxin, and IFN gamma ELISPOT responses to listeriolysin and nucleoprotein peptides.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth L Hohmann, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Eypper EH, Johnson PV, Purro EI, Hohmann EL. Transcutaneous immunization of healthy volunteers with an attenuated Listeria monocytogenes vaccine strain and cholera toxin adjuvant. Vaccine. 2013 Jul 11;31(32):3257-61. doi: 10.1016/j.vaccine.2013.05.028. Epub 2013 May 22. PMID 23707162